CLINICAL TRIAL: NCT07175246
Title: Exploring the Patterns of Sleep Disordered Breathing in Systemic Sclerosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Ahmed, resident doctor, Assiut University
Other Study IDs: Sleep-systemic-sclerosis
Record Dates: First submitted 2025-08-21; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis; Sleep-Disordered Breathing
Keywords: systemic sclerosis; Sleep Apnea; Insomnia
MeSH Terms: conditions — Scleroderma, Systemic; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Systemic sclerosis patients: Adults (18 years and older) with a confirmed diagnosis of systemic sclerosis (2013 ACR/ EULAR criteria)
  Interventions: Diagnostic Test: Polysomnography (PSG)

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) — Polysomnography (PSG) is the gold standard, multi-parametric diagnostic test used to comprehensively assess sleep architecture and diagnose sleep disorders. This objective, overnight recording captures simultaneous physiological data channels, including electroencephalography (EEG) to stage sleep, electrooculography (EOG) to detect eye movements, electromyography (EMG) to measure muscle tone, electrocardiography (ECG) for heart rhythm, respiratory effort (via thoracic and abdominal belts), nasal airflow, and pulse oximetry for blood oxygen saturation. As the primary/secondary outcome measure, PSG will be administered to quantitatively evaluate the intervention's effect on key sleep parameters such as total sleep time (TST), sleep efficiency (SE), wake after sleep onset (WASO), latency to sleep onset, and the frequency of sleep-disordered breathing events (e.g., Apnea-Hypopnea Index, AHI) or periodic limb movements.

SUMMARY:
Systemic sclerosis (SSc) is a chronic autoimmune connective tissue disease characterized by progressive fibrosis of the skin and internal organs. Fatigue, non-restorative sleep, and poor sleep quality are frequently reported among patients with SSc, yet these symptoms remain under-recognized and under-investigated in clinical practice. Despite growing awareness of the burden of sleep-related symptoms, there is a significant lack of objective data regarding sleep disturbances in this population, particularly those assessed using polysomnography (PSG).

DETAILED DESCRIPTION:
Emerging evidence suggests a notable prevalence of sleep-disordered breathing (SDB), including obstructive sleep apnea (OSA), as well as periodic limb movement disorder (PLMD) and insomnia in individuals with SSc. The multi-factorial aetiology of sleep disturbances in SSc may involve fibrotic changes in the lungs, gastroesophageal reflux, musculoskeletal discomfort, and psychological stress. Moreover, pulmonary fibrosis and restrictive lung disease in SSc have been linked to an increased risk of nocturnal hypoxia and sleep fragmentation, which may worsen fatigue and impair quality of life.

Objective sleep assessment through PSG can provide essential insights into the type and severity of sleep disorders in SSc patients. Identifying these disorders early may guide more targeted management strategies, improve patients' daily functioning, and potentially alter disease outcomes. Hence, this study is warranted to fill the existing gap in knowledge and to explore the clinical implications of sleep disturbances in systemic sclerosis.

Study Objectives is to assess the occurrence and types of sleep disorders in systemic sclerosis patients, to evaluate polysomnographic findings in systemic sclerosis disease.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years, with Confirmed diagnosed of SSc (2013 ACR/EULAR criteria).

Exclusion Criteria:

* Pre-existing primary sleep disorders diagnosed before SSc diagnosis
* Use of sedatives or hypnotics within the last month that significantly alter sleep architecture
* Severe psychiatric or neurological conditions
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years, with Confirmed diagnosed of SSc (2013 ACR/EULAR criteria)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
sleep disorders in systemic sclerosis patients | 6 hours
  Apnea-Hypopnea Index (AHI)
  Description: Average number of apneas and hypopneas per hour of sleep, assessed by overnight polysomnography.
  Unit of Measure: Events per hour
  Time Frame: 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eman Ahmed Abd Elhamed, Resident, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cholerzynska H, Zasada W, Tselios K, Grygiel-Gorniak B. Sleep Disorders in Connective Tissue Diseases-Coexisting Diseases or Disease Components? J Clin Med. 2024 Jun 22;13(13):3656. doi: 10.3390/jcm13133656. PMID 38999222
- [Background] Wongthawa N, So-Gnern A, Mahakkanukrauh A, Suwannaroj S, Foocharoen C. Sleep quality and clinical association with sleep disturbance in systemic sclerosis. BMC Rheumatol. 2023 Jul 21;7(1):21. doi: 10.1186/s41927-023-00346-7. PMID 37480089